CLINICAL TRIAL: NCT02045823
Title: Topcon 3D OCT-1 Maestro and 3D OCT-2000 Optical Coherence Tomography Systems: Agreement and Precision Study
Brief Title: OCT Agreement and Precision Study
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Maestro2000AP
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Normal Eyes; Eyes With Glaucoma; Eyes With Retinal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: Normal results from clinical exam and free of ocular pathology
- Glaucoma: Clinical exam with results consistent with glaucoma and visual field defects consistent with glaucoma
- Retina: clinical exam with results consistent with retina pathology

SUMMARY:
To demonstrate clinical substantial equivalence of 3D OCT-1 Maestro as comparable to the commercially available iVue and NW-300. Also, to demonstrate clinical substantial equivalence of 3D OCT-2000 Maestro as comparable to the commercially available NW-300.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to Criteria participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (eyes without pathology)
4. lOPs 21mmHg bilaterally
5. BCVA 20/40 or better (each eye)
6. Both eyes must be free of eye disease

Exclusion Criteria for Normal Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result abnormal, defined as GHT 'Outside Normal Limits' and/or PSD < 5%
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses> 33% or false positives> 25%, or false negatives> 25%
5. Presence of any ocular pathology except for cataract
6. Previous ocular surgery or laser treatment, other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning
7. Narrow angle
8. History of leukemia, dementia or multiple sclerosis
9. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Glaucoma Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with glaucoma
4. BCVA 20/40 or better in the study eye
5. HFA visual field (24-2 Sita Standard, white on white) result abnormal, defined as GHT 'Outside Normal Limits' and/or PSD < 5% in the study eye

Exclusion Criteria for Glaucoma Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result unreliable, defined as fixation losses> 33% or false positives> 25%, or false negatives > 25% in the study eye
4. Presence of any ocular pathology except glaucoma in the study eye
5. Previous ocular surgery or laser treatment, other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning in the study eye
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Retina Disease Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with retinal disease
4. lOP<= 21mmHg in the study eye
5. BCVA 20/400 or better in the study eye
6. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Cystoid Macula Edema, and others

Exclusion Criteria for Retinal Disease Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. Presence of glaucoma or any ocular pathology other than a Retinal pathology (e.g., cornea pathology) in the study eye
4. Previous ocular surgery or laser treatment other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning in the study eye
5. Narrow angle in the study eye
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that are Normal, or shows signs of Glaucoma, or Retinal Ocular Pathology.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sinai, PhD, Principal Investigator — Topcon Corporation
Locations (1):
- New York VA, Jamaica, New York, United States